CLINICAL TRIAL: NCT06715592
Title: Monocentric Phase II Study on the Use of Electrochemotherapy in the Treatment of Paget's Disease and High-grade Squamous Precancerous Lesions or Initially Invasive Vulvar Lesions (GinOnc-ECT Study).
Brief Title: ECT STUDY High-grade or Initially Invasive Vulva - GinOnc-ECT Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Corrado Giacomo, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GinOnc-ECT study
Record Dates: First submitted 2024-11-20; First posted 2024-12-04 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Paget Disease of the Vulva; Vulva Cancer
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Bleomycin; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECT Electrochemotherapy (Experimental): The ways in which ECT treatment will be applied have been codified at European level from the 2006 ESOPE study
  Interventions: Drug: Bleomicina

INTERVENTIONS:
Drug: Bleomicina — Colposcopically guided ECT following intralesional administration / intravenous Bleomycin or intralesional Cisplatin according to ESOPE recommendations. Reassessment after 30 days by colposcopy and conization with acquisition of histological examination.
  Other Names: CISPLATIN

SUMMARY:
Patients with a new diagnosis or recurrence of high-grade squamous precancerous lesions or initially non-invasive vulvar Paget's disease, who have not undergone other types of treatment, will be considered at the Fondazione Policlinico Universitario A. Gemelli - IRCCS - in Rome.

DETAILED DESCRIPTION:
Vulvar Paget's disease (VPD) constitutes approximately 1-2% of malignant vulvar neoplasms in its invasive form and is the most frequent localization (60%) of extramammary Paget's disease (EMPD). Due to its rarity, precise epidemiological data are not available, although the estimated incidence of EMPD in Europe is 0.7/100,000/year. The affected population is mainly comprised of postmenopausal Caucasian women. The most common clinical symptoms are vulvar itching, pain, or burning, although patients can remain asymptomatic for many years, leading to frequent diagnostic delays. Primary lesions appear as erythematous or eczematous plaques with frequent multifocal discoloration and hyperkeratosis.

The pathogenesis is not fully understood. The most accepted theories suggest a probable origin from apocrine glands, mammary-like glands, totipotent cells of the basal layer of the epidermis or cutaneous appendages, or Toker cells located at the vulvar level. From an anatomopathological point of view, it is described as an intraepithelial adenocarcinoma with apocrine or eccrine differentiation, characterized by large cells with clear cytoplasm called Paget cells. The Wilkinson and Brown classification is currently the most used, distinguishing between a primary (cutaneous) form and a secondary form associated with adenocarcinomas from other sites. Specifically, the primary form includes a type 1a intraepithelial (75-81%), type 1b invasive (16-19%), and type 1c with intraepithelial Paget cells associated with an underlying vulvar adenocarcinoma (4-17%). The secondary form is the result of pagetoid dissemination of neoplastic elements from a contiguous anorectal (type 2) or urogenital neoplasm (type 3).

The invasive primary form is characterized by a poor prognosis with a high recurrence rate and mortality (5-year survival between 0 and 15% for frankly invasive forms), and therefore, it is generally treated with extensive and demolitive surgery, complemented with radiotherapy and/or chemotherapy, with often unsatisfactory results. Even in non-invasive primary forms, the most commonly used therapeutic approach is surgical, despite the absence of clear superiority over other treatments.

Vulvar carcinoma is a rare tumor, with an incidence in Italy ranging from 0.3 to 1.8 per 100,000 population, predominantly affecting individuals aged 55 and older. Squamous cell carcinomas represent approximately 95% of vulvar carcinomas, while the remaining cases consist of melanomas, sarcomas, and basal cell carcinomas. These forms have two fundamental pathogenetic pathways, which are dependent on specific risk factors. The most frequent pathway is associated with precancerous conditions such as inflammatory epithelial diseases of the vulva. This pathway is linked to forms with an incidence in middle to advanced age (55-85 years), showing a relatively low HPV infection rate and consequently a low risk of cervical cancer. The main precancerous condition associated with the development of HPV-negative vulvar carcinoma is lichen sclerosus. Less frequently, vulvar carcinoma arises following high-risk HPV infection. This etiopathogenic pathway is more common in younger women (under 40 years), consistent with the spread of the virus.

HPV-induced carcinogenesis takes years or decades to manifest, and there is growing evidence that additional tumor-promoting stages are necessary. It is widely accepted that effective immune control is required to prevent persistent HPV infection. However, recent

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of de novo or recurrent vulvar VIN 2-3, microinvasive vulvar carcinoma in situ, and non-invasive vulvar Paget's disease
* Positivity for high-risk cervical and/or vaginal HPV
* Age > 18 years
* Karnofsky performance status >70%
* Informed consent to participate in the study
* No surgical treatment indication due to disease extension, patient refusal, anesthesiological or reconstructive reasons
* Negative Beta-hCG measurement in urine (pregnancy test or urinary beta-HCG) or in blood (plasma beta-HCG)

Exclusion Criteria:

* Patients with a histological diagnosis of adenocarcinoma
* Patients with concomitant and/or previous tumors
* Current pregnancy and breastfeeding
* Chronic renal insufficiency
* Chronic renal dysfunction
* Patients with a cardiac pacemaker
* Epilepsy
* Lung diseases with moderate/severe respiratory insufficiency
* Poor lung function or abnormal lung function
* Significant coagulation disorders
* Coagulation abnormalities (platelets < 70,000/mm³ and INR > 1.5)
* Ongoing HPV vaccination
* Patients with immunosuppressive conditions or treatments (HIV positive)
* Allergy to Bleomycin and/or Cisplatin
* Cumulative doses of 250 mg/m² of Bleomycin received

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the activity of electrochemotherapy in the treatment of vulvar lesions and noninvasive M. of Paget | 30 days post treatment and then Outpatient visit at 3, 6 and 12 months from procedures.
  Evaluation of treatment response will be done by histological analysis of surgical specimens after lesion excision at 30 days after ECT.Thereafter, patients will be evaluated by the gynecologic oncologist in the outpatient clinic at 3,6 and 12 months after the procedure.Inspection of the genitals and pelvic region will be performed during the follow-ups,and if necessary,new biopsies of the previously treated area will be taken.Criteria for response to ECT will be defined as:complete response(CR)when there is disappearance of the pre-tumor/tumor lesion;partial response(PR )if the lesion appears reduced by more than 30% in the product between the two major perpendicular diameters; stable disease(NC=no change)when the lesion is reduced by less than 30% or increased by less than 20% of its volume;disease progression(PD)if there is a lesion size increase of at least 20%.In cases where it is not objectively possible to measure tumor size,the response will be recorded as "not evaluable"(NV).

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Corrado, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Lazio, Italy